CLINICAL TRIAL: NCT01121562
Title: A Phase II Study Of Sunitinib In Patients With Progressive Advanced/Metastatic Well-Differentiated Pancreatic Neuroendocrine Tumors
Brief Title: Efficacy And Safety Of Sunitinib In Patients With Advanced Well-Differentiated Pancreatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181193
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Pancreatic Neuroendocrine Tumors
Keywords: Neuroendocrine tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib arm (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib capsule will be given orally at continuous daily dosing with a dose of 37.5 mg in the morning (regardless fasting or non-fasting, One cycle will be 28days)

SUMMARY:
The purpose of the study is to evaluate the effect of Sunitinib on the clinical benefit response rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced (unresectable or metastatic) biopsy-proven pancreatic NET (Neuroendocrine Tumor)

Exclusion Criteria:

* Patients with poorly differentiated neuroendocrine cancer are not eligible

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Japan (4):
  - Aichi Cancer Center Central Hospital, Nagoya, Aichi-ken
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Osaka Police Hospital, Osaka, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo

REFERENCES:
- [Derived] Ito T, Okusaka T, Nishida T, Yamao K, Igarashi H, Morizane C, Kondo S, Mizuno N, Hara K, Sawaki A, Hashigaki S, Kimura N, Murakami M, Ohki E, Chao RC, Imamura M. Phase II study of sunitinib in Japanese patients with unresectable or metastatic, well-differentiated pancreatic neuroendocrine tumor. Invest New Drugs. 2013 Oct;31(5):1265-74. doi: 10.1007/s10637-012-9910-y. Epub 2012 Dec 27. PMID 23269537
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181193&StudyName=Efficacy%20And%20Safety%20Of%20Sunitinib%20In%20Patients%20With%20Advanced%20Well-Differentiated%20Pancreatic%20Neuroendocrine%20Tumors

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: Sunitinib 37.5 mg was orally administered once daily in a continuous daily dosing regimen (1 cycle = 4 weeks).
Period: Overall Study
Arm/Group | Sunitinib
Started | 12
Completed | 0
Not Completed | 12
Not completed — Objective progression or relapse | 8
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Sponsor Decision | 1
Not completed — Met study discontinuation criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Response Rate (CBR)
Description: CBR rate is defined as the percentage of participants with a best overall response of confirmed complete response (CR), confirmed partial response (PR) ,or stable disease (SD) ≥ 24 weeks.
  Based on RECIST, CR is defined as the disappearance of all target lesions and PR is defined as a greater than or equal to 30% decrease in the sum of the longest dimensions of the target lesion. SD is defined neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest dimensions since the treatment started.
Time Frame: Up to 799 days of treatment
Population: Full Analysis Set was defined as the population of all enrolled participants in whom well-differentiated pancreatic neuroendocrine tumor had been diagnosed and who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 12
percentage of participants | 75.0 [42.8 to 94.5]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response of confirmed CR or confirmed PR. Based on the response evaluation criteria in solid tumors (RECIST), CR is defined as the disappearance of all target lesions and PR is defined as a greater than or equal to 30% decrease in the sum of the longest dimensions of the target lesion.
Time Frame: Up to 799 days of treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 12
percentage of participants | 50.0 [21.1 to 78.9]

3. Secondary Outcome: Tumor Shrinkage
Description: Tumor shrinkage is defined as the percent change from baseline for the sum of the longest diameter of target lesions in participants.
Time Frame: Up to 799 days of treatment
Population: Full Analysis Set was defined as the population of all enrolled participants in whom well-differentiated pancreatic neuroendocrine tumor had been diagnosed and who received at least one dose of study medication. "n " in the measured values means number of participants analyzed in the cycle.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sunitinib
Number analyzed (Participants) | 12
percent change
  Cycle 1 (n=1) | -20.0 (NA) — Only 1 participant was analyzed in this cycle
  Cycle 2 (n=11) | -14.4 (13.43)
  Cycle 3 (n=12) | -18.0 (17.70)
  Cycle 5 (n=9) | -26.0 (10.03)
  Cycle 7 (n=9) | -28.5 (11.86)
  Cycle 9 (n=9) | -31.8 (17.20)
  Cycle 11 (n=9) | -36.4 (30.11)
  Cycle 13 (n=9) | -28.8 (16.92)
  Cycle 14 (n=1) | 1.7 (NA) — Only 1 participant was analyzed in this cycle
  Cycle 15 (n=7) | -32.5 (17.29)
  Cycle 16 (n=1) | -34.7 (NA) — Only 1 participant was analyzed in this cycle
  Cycle 17 (n=5) | -38.7 (15.41)
  Cycle 18 (n=1) | -43.1 (NA) — Only 1 participant was analyzed in this cycle
  Cycle 19 (n=4) | -37.8 (19.21)
  Cycle 21 (n=4) | -35.8 (19.19)
  Cycle 23 (n=4) | -35.1 (22.82)
  Cycle 25 (n=4) | -32.6 (19.64)
  Cycle 27 (n=3) | -30.8 (26.68)
  Cycle 28 (n=2) | -40.4 (9.72)
  Cycle 29 (n=1) | 3.3 (NA) — Only 1 participant was analyzed in this cycle
  Maximum Reduction (n=12) | -34.8 (28.76)

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from registration to first documentation of progressive disease (PD) or to death due to any cause, whichever occurs first.
Time Frame: Up to 799 days of treatment
Population: Full Analysis Set was defined as the population of all enrolled participants in whom well-differentiated pancreatic neuroendocrine tumor had been diagnosed and who received at least one dose of study medication.
  Median PFS had not yet been reached due to short of events.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 12
Months | 16.8 [9.3 to 26.2]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from registration to documentation of death due to any cause.
Time Frame: Up to 3 years from the last subject registration to the study
Population: Full Analysis Set was defined as the population of all enrolled participants in whom well-differentiated pancreatic neuroendocrine tumor had been diagnosed and who received at least one dose of study medication.
  OS was not analyzed due to short of events.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 12
Months | NA [22.0 to NA] — Median OS had not yet been reached due to short of events.

6. Secondary Outcome: Dose-corrected Trough Plasma Concentrations of Sunitinib, SU012662 and Total Drug (Sunitinib + SU012662).
Description: Reference dose is 37.5 mg. Dose-corrected concentration is calculated from the following formula, "observed concentration multiplied by 37.5" over "actual dose".
  SU012662 is an active metabolite of sunitinib.
Time Frame: Predose of Cycle 1 Day15, Cycle 2 Day1, Cycle 3 Day1, and Cycle 4 Day 1
Population: The pharmacokinetics analysis set was defined as all participants who had at least one plasma concentration data at trough sampling with steady-state condition. "n" in the measured values means number of participants analyzed.
Measure: Mean (Standard Deviation); unit: nanogram/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 11
nanogram/mL
  Sunitinib (Cycle 1 Day 15, n=10) | 53.9 (17.6)
  Sunitinib (Cycle 2 Day 1, n=2) | 41.7 (21.9)
  Sunitinib (Cycle 3 Day 1, n=8) | 49.9 (19.7)
  Sunitinib (Cycle 4 Day 1, n=5) | 53.5 (24.6)
  SU012662 (Cycle 1 Day 15, n=10) | 23.7 (7.00)
  SU012662 (Cycle 2 Day 1, n=2) | 21.2 (6.36)
  SU012662 (Cycle 3 Day 1, n=8) | 25.7 (9.14)
  SU012662 (Cycle 4 Day 1, n=5) | 19.6 (7.44)
  Total drug (Cycle 1 Day 15, n=10) | 77.5 (20.9)
  Total drug (Cycle 2 Day 1, n=2) | 62.9 (28.3)
  Total drug (Cycle 3 Day 1, n=8) | 75.5 (26.5)
  Total drug (Cycle 4 Day 1, n=5) | 73.0 (28.8)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=12)
Enterocolitis (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Convulsion (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=12)
Anaemia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 2
Hypothyroidism (Endocrine disorders) | 4
Conjunctival haemorrhage (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Eyelash discolouration (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 2
Glossitis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Loose tooth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Oral dysaesthesia (Gastrointestinal disorders) | 2
Periodontitis (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Face oedema (General disorders) | 1
Fatigue (General disorders) | 7
Malaise (General disorders) | 2
Mucosal inflammation (General disorders) | 3
Oedema (General disorders) | 4
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 5
Cholangitis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Encephalitis herpes (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Infected epidermal cyst (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 5
Oral herpes (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyoderma (Infections and infestations) | 1
Skin candida (Infections and infestations) | 1
Trichophytosis (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood urine present (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 1
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 2
Protein urine present (Investigations) | 2
Urine output decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysaesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 7
Hypoaesthesia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Scrotal haematocoele (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.